CLINICAL TRIAL: NCT00563407
Title: Novel Surrogate Markers as Predictors of Radiation Toxicity in Breast Cancer Patients Undergoing Helical Tomotherapy Compared to Standard Radiation Therapy
Status: Terminated | Type: Observational
Why Stopped: accrual goal met
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: BR-1-0090
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2011-09

CONDITIONS: Genetic Markers; Cardiac Toxicity; Breast and Skin Motion
Keywords: skin toxicity prediction; cardiac toxicity prediction
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Radiotherapy is standard treatment for breast cancer after lumpectomy. Although this treatment showed substantial patient benefits and decrease of local recurrence and deaths from breast cancer, it also results in some severe late side-effects, such as skin fibrosis and cardiac failure. It's possible to offer breast irradiation (RT) and minimizing toxicities radiation dose to skin, lung and heart. This will be achieved with highly conformal RT delivery using Tomotherapy. We plan to evaluate this approach in clinical study. We plan also to evaluate the value of genomic, cellular and functional imaging endpoints as predictive markers of toxicity in our breast cancer population. This program is expected to prospectively validate that Tomotherapy for breast RT can decrease skin, lung and heart toxicities and maintaining excellent cancer control after lumpectomy.

DETAILED DESCRIPTION:
Radiotherapy is standard treatment after conservative surgery for early-stage breast cancer. Although this approach substantially improves local control and reduces deaths from breast cancer, it also results in some severe late side-effects, including skin fibrosis, deaths from radiation-induced cardiac disease and lung cancer. We will undertake a novel approach to the evaluation of radiation-induced toxicity during and after whole breast irradiation (RT) following breast-conserving surgery, with the long-term strategic goal of minimizing RT toxicity in early breast cancer. Theoretically, it is possible to achieve this goal through very highly conformal RT delivery and avoidance of RT in toxicity-prone individuals where possible. We plan to evaluate the utility of genomic analysis, cellular DNA repair competence, and functional imaging endpoints as predictive markers of toxicity in our breast cancer population. This program is expected to (a) prospectively validate that HT for breast RT can decrease acute toxicity whilst maintaining excellent cancer control after BCS; (b) demonstrate that novel surrogate markers will aid in the prediction of acute and/or late normal tissue toxicity with a view to identify toxicity-prone (or conversely, robust) individuals from amongst the breast cancer population.

ELIGIBILITY:
Inclusion Criteria:

* early breast cancer treated with lumpectomy
* must have T1-2 N0-1 invasive carcinoma of the breast
* must sign an informed consent
* must be at least 18 years of age

Exclusion Criteria:

* collagen vascular disease
* metastatic disease
* pregnant or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with early breast cancer (carcinoma insitu , T1-2, N0-1) treated with lumpectomy.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2006-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
skin and cardiac toxicity | 24 months post RT

SECONDARY OUTCOMES:
prediction | 24 months post RT

CONTACTS AND LOCATIONS:
Overall Officials: Bassam Abdulkarim, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Alberta Cancer Board, Edmonton, Alberta, Canada